CLINICAL TRIAL: NCT07072286
Title: RELIEVED (REgionaL anesthesIa PElVic fracturEs stuDy) Study. Regional Anesthesia (RA) Techniques for Pain Management in Pelvic Fractures: A Prospective, Monocentric, Pilot Cohort Study. Pain Management in Surgical and Conservative Settings."
Brief Title: RELIEVED (REgionaL anesthesIa PElVic fracturEs stuDy) Study. Regional Anesthesia (RA) Techniques for Pain Management in Pelvic Fractures: A Prospective, Monocentric, Pilot Cohort Study.
Acronym: RELIEVED
Status: Recruiting | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Sponsor
Other Study IDs: 00179/2024
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Bone Injury; Pelvis Injury; Acetabular Fractures; Acetabular Surgery; Trauma Injury
Keywords: regional anethesia; pain management; pelvic fractures; acetabular fractures; surgery
MeSH Terms: conditions — Accidental Injuries; Agnosia; Hip Fractures | interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA group: Patients treated with RA techniques in association to multimodal analgesia
  Interventions: Procedure: Regional Anesthesia; Drug: Multimodal analgesia
- Multimodal Analgesia Group: Patients treated with multimodal analgesia alone
  Interventions: Drug: Multimodal analgesia

INTERVENTIONS:
Procedure: Regional Anesthesia — * Supra-inguinal fascia iliaca block (SIFI)
  * Lumbar erector spinae plane block (ESP)
  * Transmuscular quadratus lumborum block (QLB) All blocks will be performed by experienced anesthesiologists under ultrasound guidance, using long-acting anesthetics (ropivacaine) at fixed concentrations and doses within weight-based safety limits.
  Groups: RA group
Drug: Multimodal analgesia — All enrolled subjects will be treated according to the standard analgesic protocol for pelvic fractures, in accordance with available literature and institutional guidelines. Specifically, the protocols include the use of multimodal analgesia techniques in line with current clinical practice, including paracetamol, non-steroidal anti-inflammatory drugs, opioids.

SUMMARY:
The goal of this observational clinical trial is to assess the impact of Regional Anesthesia (RA) techniques with the strongest anatomical and scientific support in controlling acute post-operative pain in pelvic/acetabular fractures, as well as their potential role in reducing complications related to excessive intra- and postoperative opioid use.

The main questions it aims to answer are:

Does RA lower opioid use in the first 24 hours after pelvic/acetabular fractures surgery? Does RA lower pain scores in the first 48 hours after surgery, incidence of complications and occurrence of persistent post-surgical pain?

During the hours and days following surgery, the research team will evaluate and assess the intensity of any postoperative pain at predefined time points; quantify the use of pain medications and any related complications; and measure the possible onset of chronic pain and the timeline of functional recovery (through scheduled clinical follow-up at 30, 60, and 90 days).

Participants will:

at the time of surgery, and only in the presence of trained and certified anesthesiologists, patients will receive regional anesthesia techniques in addition to the standard multimodal analgesic treatment. In the absence of certified anesthesiologists, patients will be treated exclusively with systemic multimodal analgesia according to the standard protocol.

All the procedures are part of the current clinical practice and no experimental techniques or medications are involved.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ability to provide informed consent
* Patients with pelvic/acetabular fractures requiring surgery

Exclusion Criteria

* Age < 18 years
* Absolute contraindications to ALR techniques (uncorrectable coagulopathies, known allergy to local anesthetics, technical impossibility of execution)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pelvic/acetabular fractures presenting to the Emergency and Trauma Department, either as primary transport or secondary referral, who require surgery (percutaneous or via open reduction/internal fixation).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-07-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | Up to 24 hours after surgery
  Post-operative opioid consumption (morphine milligram equivalents - MMEs) in the first 24 hours.

SECONDARY OUTCOMES:
Pain Scores | post-operatively at 6, 12, 24 and 48 hours following surgery
  Area under the curve (AUC) of acute pain scores (measured via Numeric Rating Scale - NRS)
Persistent post-surgical pain | 30, 60, 90-days after surgery
  Incidence of chronic post-operative/post-traumatic pain assessed via Numeric rating scale (NRS) through telephone follow-up.
Opioids Side Effects | Up to 48 hours after surgery
  Incidence of acute side effects related to opioid use (excessive sedation, nausea/vomiting, respiratory depression, pruritus, urinary retention, constipation).
RA side effects | Up to 48 hours after surgery
  Incidence of complications related to nerve blocks (block failure, nerve damage, hematoma, systemic local anesthetic toxicity).
Hospital length of stay | From surgery up to the first follow up at 30 days
  Days of admission in the hospital where surgery is provided

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Traumatologico Ortopedico (CTO) - AOU Città della Salute e della Scienza Univeristy Hospital, Turin, Italy

IPD SHARING:
Plan to Share IPD: Undecided